CLINICAL TRIAL: NCT02160392
Title: Virologic, Pharmacologic, and Immunologic Characterization of the Female Upper Genital Tract in HIV-infected Women
Brief Title: Female Upper Genital Tract in HIV-infected Women
Acronym: FUGTS
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Lisa Rahangdale, MD, MPH, Assistant Professor, University of North Carolina, Chapel Hill
Other Study IDs: FUGTS2010
Record Dates: First submitted 2014-06-05; First posted 2014-06-10 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: HIV
Keywords: HIV; female; genital tract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Endometrial and cervical lavage specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Endometrial biopsy: HIV + and HIV negative women underwent lower and upper genital tract sampling.
  Interventions: Procedure: Endometrial biopsy

INTERVENTIONS:
Procedure: Endometrial biopsy — Endometrial biopsy (EMB) specimens were collected via a 3 mm diameter plastic pipelle that was inserted into the uterus following EML. A sample of tissue was obtained by retracting the pipelle's plunger leading to negative suction and rotating the cannula for approximately 15 seconds.

SUMMARY:
The female upper genital tract is a unique compartment involved in HIV pathogenesis.

DETAILED DESCRIPTION:
The persistent detection of HIV in the female genital tract in spite of ART is unexplained, and it is possible the uterine endometrium serve as a reservoir. There are limited data regarding the interaction between HIV expression, antiretroviral therapy (ART) and host immune system in the uterine endometrium.

ELIGIBILITY:
Inclusion Criteria:

* Regularly menstruating women (between 21-42 days)
* between ages 25-50 years
* Fully suppressed by antiretroviral therapy with plasma HIV RNA < 40 copies/mL within the last 6 months.

Exclusion Criteria:

* Pregnant or planning pregnancy
* Unwilling to use 2 forms of contraception (condoms + hormonal) if they did not have previous bilateral tubal ligation procedure
* Intrauterine device in place
* Untreated cervical infection (N. gonnorhea, C. trachomatis)
* Taking immunosuppressive medications

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We enrolled HIV-1 positive menstruating women between ages 25-48 years.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2010-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Immune characteristics | Single visit approximately 14-42 days after the first day of the last menstrual period.
  Endometrial lavage (EML) and biopsy (EMB) samples were compared to cervicovaginal lavage (CVL) and fluid (CVF) samples from HIV-negative healthy women (N=x) and HIV-infected women (n=x) taking ART with plasma HIV RNA <40 copies/mL. All participants were in the luteal phase of the menstrual cycle. Immunologic study was completed using Luminex and flow cytometry. Concentrations of tenofovir (TFV), emtricitabine (FTC) and their active intracellular metabolites (TFVdp and FTCtp) were measured using LC-MS/MS in 11 HIV-infected women. HIV RNA was measured in plasma, EML and CVL using the Abbott RealTime HIV-1 assay (lower limit of detection 40 copies/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Rahangdale, MD, MPH, Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC, Chapel Hill, North Carolina, United States